CLINICAL TRIAL: NCT03522077
Title: RAVE: Radial Artery Vascular Complication and Resource Utilization in Subjects Undergoing an Angiogram/PCI (Percutaneous Coronary Intervention)
Brief Title: RAVE: Radial Artery Vascular Complication and Resource Utilization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Chitogen, Inc. (Individual)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00106906; 17-132 (Other: Aurora St Lukes Medical Center)
Record Dates: First submitted 2018-04-30; First posted 2018-05-11 (Actual); Results first posted 2023-02-09 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2023-01

CONDITIONS: Angiogram; Percutaneous Coronary Intervention
Keywords: Angiogram; Hemostatic; Activated clotting time; Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- RadAR EasyCLik plus SoftSeal®-STF hemostatic pad (Experimental): Hemostasis will be obtained with the SoftSeal®-STF hemostatic pad and vascular compression device by applying pressure at the point proximal and distal to the puncture site and removing the sheath. While still maintaining pressure, the SoftSeal®-STF hemostatic pad will be applied over the puncture site. The cath lab staff will allow a small amount of blood (< 0.2 mL) to contact the surface of the hemostatic pad and then will apply constant pressure with a vascular compression device.
  Interventions: Device: RadAR EasyCLik plus ®-STF hemostatic pad
- TR BAND® plus SoftSeal®-STF hemostatic pad (Active Comparator): Hemostasis will be obtained with the SoftSeal®-STF hemostatic pad and vascular compression device by applying pressure at the point proximal and distal to the puncture site and removing the sheath. While still maintaining pressure, the SoftSeal®-STF hemostatic pad will be applied over the puncture site. The cath lab staff will allow a small amount of blood (< 0.2 mL) to contact the surface of the hemostatic pad and then will apply constant pressure with a vascular compression device.
  Interventions: Device: TR BAND® Compression device plus ®-STF hemostatic pad
- SoftSeal®-STF hemostatic (Experimental): Hemostasis at the radial access site for subjects randomized to the SoftSeal®-STF hemostatic pad will be obtained by applying pressure at the point proximal and distal to the puncture site and removing the sheath. While still maintaining pressure, the SoftSeal®-STF hemostatic pad will be applied over the puncture site. The cath lab staff will allow a small amount of blood (< 0.2 mL) to contact the surface of the hemostatic pad and then will apply constant pressure.
  Interventions: Device: SoftSeal®-STF hemostatic pad
- VascBand™ Hemostat (Active Comparator): Hemostasis at the radial access for subjects randomized to the VascBand™ Hemostat will be obtained in accordance to the manufacturer's instructions. The VascBand™ device will be placed proximal to the puncture site and inflated slowly while simultaneously removing the sheath, and continue to inject air (max. 18 mL) into the device until hemostasis is obtained.
  Interventions: Device: VascBand™ Hemostat

INTERVENTIONS:
Device: RadAR EasyCLik plus ®-STF hemostatic pad — Chitosan-based, non-woven pad with a unique, proprietary fiber structure that when hydrated with tissue fluids forms a gel-like synthetic clot in conjunction with the RadAR EasyCLik compression device
  Arms: RadAR EasyCLik plus SoftSeal®-STF hemostatic pad
Device: TR BAND® Compression device plus ®-STF hemostatic pad — Chitosan-based, non-woven pad with a unique, proprietary fiber structure that when hydrated with tissue fluids forms a gel-like synthetic clot in conjunction with the TR BAND® compression device
  Arms: TR BAND® plus SoftSeal®-STF hemostatic pad
Device: SoftSeal®-STF hemostatic pad — Chitosan-based, non-woven pad with a unique, proprietary fiber structure that when hydrated with tissue fluids forms a gel-like synthetic clot
  Arms: SoftSeal®-STF hemostatic
Device: VascBand™ Hemostat — The VascBand™ Hemostat is an FDA-approved compression device designed to assist hemostasis of arterial, venous and hemodialysis percutaneous access sites.
  Arms: VascBand™ Hemostat

SUMMARY:
The primary objective of this study is to determine if there is a reduction in time to hemostasis in subjects treated with SoftSeal®-STF hemostatic pad when used in conjunction with a vascular compression device after radial transcatheter procedure.

DETAILED DESCRIPTION:
The SoftSeal-STF hemostatic pad and compression devices (TR BAND® and RadAR EasyCLik) function to stop bleeding without obstructing radial artery flow, and have been shown to reduce the occurrence of radial artery occlusion.

The SoftSeal-STF hemostatic pad is an FDA-approved, chitosan-based, non-woven pad with a unique, proprietary fiber structure that when hydrated with tissue fluids forms a gel-like synthetic clot. Its mechanism of action is believed to be due to bioadhesion between the chitosan polymer chains, which are positively charged, and the negatively charged blood and tissue components, thereby stopping bleeding.

In this study the RadAR EasyCLik and TR BAND® Compression devices will be used with the SoftSeal®-STF hemostatic pad to promote hemostasis at the puncture site. Both vascular compression devices are FDA approved.

The VascBand™ Hemostat is an FDA-approved compression device designed to assist hemostasis of arterial, venous and hemodialysis percutaneous access sites.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for an angiogram/PCI
* Planned transradial approach

Exclusion Criteria:

* Evidence of impaired dual perfusion to the hand when tested using Allen's test
* Inaccessible radial arteries due to anatomic variations
* Infection or other skin disorder at the puncture site
* Undergoing an emergent or unplanned angiogram using the transradial approach
* Evidence of severe cognitive impairment or inability to understand the study procedures and answer follow-up questions
* Known sensitivity or allergic reaction to materials in the study devices
* Unwilling to participate in the study and follow all study-related procedures
* Participating physician deems the subject to not be a good candidate
* Inability to achieve radial access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad F Jan, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Aurora Health Care, Milwaukee, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SoftSeal®-STF Hemostatic | VascBand™ Hemostat | RadAR EasyCLik Plus SoftSeal®-STF Hemostatic Pad | TR BAND® Plus SoftSeal®-STF Hemostatic Pad
Started | 49 | 51 | 100 | 100
Completed | 49 | 51 | 100 | 100
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SoftSeal®-STF Hemostatic | VascBand™ Hemostat | RadAR EasyCLik Plus SoftSeal®-STF Hemostatic Pad | TR BAND® Plus SoftSeal®-STF Hemostatic Pad | Total
Number analyzed (Participants) | 49 | 51 | 100 | 100 | 300
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 66 [58 to 72] | 65 [58 to 71] | 68 [58 to 74] | 65 [58 to 72] | 66 [58 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 18 | 34 | 41 | 117
  Male | 25 | 33 | 66 | 59 | 183
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2 | 5 | 9
  Not Hispanic or Latino | 48 | 50 | 98 | 95 | 291
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  Black or African American | 6 | 7 | 11 | 14 | 38
  White | 43 | 43 | 88 | 86 | 260
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Hypertension [Count of Participants; unit: Participants] | 40 | 45 | 83 | 86 | 254

OUTCOME MEASURES:

1. Primary Outcome: Time to Hemostasis
Description: Time interval in minutes beginning with sheath removal and ending with removal of hemostatic device and/or observed hemostasis
Time Frame: 1 day
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | SoftSeal®-STF Hemostatic | VascBand™ Hemostat | RadAR EasyCLik Plus SoftSeal®-STF Hemostatic Pad | TR BAND® Plus SoftSeal®-STF Hemostatic Pad
Number analyzed (Participants) | 49 | 51 | 100 | 100
minutes | 19 [15 to 30] | 120 [120 to 124] | 44 [40 to 58.5] | 45 [40 to 69]

2. Secondary Outcome: Number of Participants With Major Access Site Bleeding
Description: A ≥ 3 mg/dL drop in hemoglobin, or required blood transfusion or vascular repair to control bleeding. Prior to discharge.
Time Frame: Post procedure to prior to discharge, on average same day discharge or up to 1-2 days
Measure: Count of Participants; unit: Participants
Arm/Group | SoftSeal®-STF Hemostatic | VascBand™ Hemostat | RadAR EasyCLik Plus SoftSeal®-STF Hemostatic Pad | TR BAND® Plus SoftSeal®-STF Hemostatic Pad
Number analyzed (Participants) | 49 | 51 | 100 | 100
Participants | 0 | 0 | 0 | 0

3. Secondary Outcome: Number of Participants With Minor Access Site Bleeding
Description: Number of participants with light access site bleeding without hematoma formation
Time Frame: Post procedure to prior to discharge, on average same day discharge or up to 1-2 days
Measure: Count of Participants; unit: Participants
Arm/Group | SoftSeal®-STF Hemostatic | VascBand™ Hemostat | RadAR EasyCLik Plus SoftSeal®-STF Hemostatic Pad | TR BAND® Plus SoftSeal®-STF Hemostatic Pad
Number analyzed (Participants) | 49 | 51 | 100 | 100
Participants | 4 | 1 | 12 | 20

4. Secondary Outcome: Number of Participants With Minor Access Site Bleeding
Description: Number of participants with light access site bleeding without hematoma formation
Time Frame: At time of follow up office visit, if done within 45 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | SoftSeal®-STF Hemostatic | VascBand™ Hemostat | RadAR EasyCLik Plus SoftSeal®-STF Hemostatic Pad | TR BAND® Plus SoftSeal®-STF Hemostatic Pad
Number analyzed (Participants) | 49 | 51 | 100 | 100
Participants | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Hematoma Formation
Description: Number of participants with hematoma formation ≥ 3 cm in diameter
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | SoftSeal®-STF Hemostatic | VascBand™ Hemostat | RadAR EasyCLik Plus SoftSeal®-STF Hemostatic Pad | TR BAND® Plus SoftSeal®-STF Hemostatic Pad
Number analyzed (Participants) | 49 | 51 | 100 | 100
Participants | 4 | 0 | 2 | 5

6. Secondary Outcome: Visual Analogue Scale (VAS)
Description: Pain at access site on numeric scale of 0-10, 0 meaning no pain at all and 10 meaning extreme pain. A lower score is a better outcome and higher score is a worse outcome.
Time Frame: 3 day
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SoftSeal®-STF Hemostatic | VascBand™ Hemostat | RadAR EasyCLik Plus SoftSeal®-STF Hemostatic Pad | TR BAND® Plus SoftSeal®-STF Hemostatic Pad
Number analyzed (Participants) | 48 | 47 | 100 | 100
score on a scale | 0.94 (1.80) | 0.51 (1.29) | 0.38 (1.31) | 0.42 (1.27)

7. Secondary Outcome: Visual Analogue Scale (VAS)
Description: as for outcome 6
Time Frame: At time of follow up office visit, if done within 45 days post procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SoftSeal®-STF Hemostatic | VascBand™ Hemostat | RadAR EasyCLik Plus SoftSeal®-STF Hemostatic Pad | TR BAND® Plus SoftSeal®-STF Hemostatic Pad
Number analyzed (Participants) | 46 | 48 | 99 | 100
score on a scale | 0.09 (0.35) | 0 (0) | 0 (0) | 0.03 (0.22)

8. Secondary Outcome: Number of Participants With Evidence of Hand/Digit Ischemia
Description: Reported as pain, tingling, or numbness in the hand and/or fingers reported
Time Frame: 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | SoftSeal®-STF Hemostatic | VascBand™ Hemostat | RadAR EasyCLik Plus SoftSeal®-STF Hemostatic Pad | TR BAND® Plus SoftSeal®-STF Hemostatic Pad
Number analyzed (Participants) | 49 | 51 | 100 | 100
Participants | 2 | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Evidence of Hand/Digit Ischemia
Description: Reported as pain, tingling, or numbness in the hand and/or fingers reported
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | SoftSeal®-STF Hemostatic | VascBand™ Hemostat | RadAR EasyCLik Plus SoftSeal®-STF Hemostatic Pad | TR BAND® Plus SoftSeal®-STF Hemostatic Pad
Number analyzed (Participants) | 49 | 51 | 100 | 100
Participants | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Participants Who Had a Readmission
Description: Number of Participants who had a Readmission for a Vascular complication
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | SoftSeal®-STF Hemostatic | VascBand™ Hemostat | RadAR EasyCLik Plus SoftSeal®-STF Hemostatic Pad | TR BAND® Plus SoftSeal®-STF Hemostatic Pad
Number analyzed (Participants) | 49 | 51 | 100 | 100
Participants | 0 | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Bruising, Swelling, or Redness
Description: Number of participants with bruising, swelling, or redness at or near access site
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | SoftSeal®-STF Hemostatic | VascBand™ Hemostat | RadAR EasyCLik Plus SoftSeal®-STF Hemostatic Pad | TR BAND® Plus SoftSeal®-STF Hemostatic Pad
Number analyzed (Participants) | 49 | 51 | 100 | 100
Participants | 5 | 3 | 5 | 6

12. Secondary Outcome: Number of Participants Who Completed Patient Satisfaction Assessment
Description: Reported as average, above average, or excellent satisfaction with procedure
Time Frame: At time of follow up office visit, if done within 45 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | SoftSeal®-STF Hemostatic | VascBand™ Hemostat | RadAR EasyCLik Plus SoftSeal®-STF Hemostatic Pad | TR BAND® Plus SoftSeal®-STF Hemostatic Pad
Number analyzed (Participants) | 49 | 51 | 100 | 100
Participants
  Average | 3 | 1 | 4 | 4
  Above average | 9 | 6 | 34 | 20
  Excellent | 33 | 41 | 60 | 76
  No response | 4 | 3 | 2 | 0

13. Secondary Outcome: Number of Participants With Level of Post Procedure Healing
Description: Satisfaction with healing post procedure, reported as average, above average, or excellent
Time Frame: At time of follow up office visit, if done within 45 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | SoftSeal®-STF Hemostatic | VascBand™ Hemostat | RadAR EasyCLik Plus SoftSeal®-STF Hemostatic Pad | TR BAND® Plus SoftSeal®-STF Hemostatic Pad
Number analyzed (Participants) | 49 | 51 | 100 | 100
Participants
  Average | 4 | 2 | 4 | 4
  Above average | 6 | 5 | 30 | 23
  Excellent | 35 | 41 | 64 | 73
  No response | 4 | 3 | 2 | 0

ADVERSE EVENTS:
Time Frame: Post procedure (considered time after procedure and prior to discharge), discharge (considered at time of discharge), 3 day follow up, and 30-45 day follow up office visit
Arm/Group | SoftSeal®-STF Hemostatic | VascBand™ Hemostat | RadAR EasyCLik Plus SoftSeal®-STF Hemostatic Pad | TR BAND® Plus SoftSeal®-STF Hemostatic Pad
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/51 | 0/100 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/51 | 0/100 | 2/100
Other Adverse Events (participants affected / at risk) | 11/49 | 1/51 | 13/100 | 15/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SoftSeal®-STF Hemostatic (N=49) | VascBand™ Hemostat (N=51) | RadAR EasyCLik Plus SoftSeal®-STF Hemostatic Pad (N=100) | TR BAND® Plus SoftSeal®-STF Hemostatic Pad (N=100)
acute frontal intraparenchymal hemorrhage. (Vascular disorders) | 0 | 0 | 0 | 1
Hematoma causing hospitalization (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SoftSeal®-STF Hemostatic (N=49) | VascBand™ Hemostat (N=51) | RadAR EasyCLik Plus SoftSeal®-STF Hemostatic Pad (N=100) | TR BAND® Plus SoftSeal®-STF Hemostatic Pad (N=100)
Minor Bleeding (Surgical and medical procedures) | 7 | 1 | 11 | 11
Hematoma (Surgical and medical procedures) | 4 | 0 | 2 | 4

LIMITATIONS AND CAVEATS:
The limitations of our study are that only the first phase of the study was randomized. The second phase was nonrandomized, which could potentially cause bias in our study. However, we used a consecutive enrollment approach where the first 100 patients were scheduled for the SoftSeal + EasyClick approach, and the subsequent 100 patients were enrolled for SoftSeal + TR Band approach.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-11): https://cdn.clinicaltrials.gov/large-docs/77/NCT03522077/Prot_SAP_000.pdf